CLINICAL TRIAL: NCT02860234
Title: Tailored Operative or Non-operative Management for MRI Defined Low-risk Rectal Cancer Following Neoadjuvant Intensity Modulated Radiotherapy With Concurrent Capecitabine Plus Consolidation CapeOX.
Brief Title: Tailored Operative or Non-operative Management for Low-risk Rectal Cancer After Intensive Neoadjuvant Treatment
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Aiwen Wu, Chief, Unit III & Ostomy Service, Gastrointestinal Cancer Center, Peking University Cancer Hospital & Institute
Other Study IDs: PKUCH-R01
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; neoadjuvant; radiotherapy; chemotherapy; organ preservation
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Radiotherapy, Intensity-Modulated; Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Group A:Clinical complete response (cCR): Patients who achieve cCR when restaged by DRE-Endoscopy-MRI-CEA at 16 weeks following intensity modulated radiotherapy(IMRT) plus consolidation CapeOX(Capecitabine+Oxaliplatin) will receive Nonoperative Management(NOM).
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: intensity modulated radiotherapy; Procedure: DRE-Endoscopy-MRI-CEA; Procedure: Nonoperative Management; Behavioral: Quality of Life Questionnaires
- Group B:Near-cCR: Patients who achieve near-cCR when restaged by DRE-Endoscopy-MRI-CEA at 16 weeks following intensity modulated radiotherapy(IMRT) plus consolidation CapeOX(Capecitabine+Oxaliplatin) will receive Local Excision(LE) or Nonoperative Management(NOM).
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: intensity modulated radiotherapy; Procedure: DRE-Endoscopy-MRI-CEA; Procedure: Nonoperative Management; Procedure: Local Excision; Behavioral: Quality of Life Questionnaires
- Group C:Residual tumor: Patients with residual tumor when restaged by DRE-Endoscopy-MRI-CEA at 16 weeks following intensity modulated radiotherapy(IMRT) plus consolidation CapeOX(Capecitabine+Oxaliplatin) will receive Total Mesorectal Excision(TME).
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: intensity modulated radiotherapy; Procedure: DRE-Endoscopy-MRI-CEA; Procedure: Total Mesorectal Excision; Behavioral: Quality of Life Questionnaires

INTERVENTIONS:
Drug: Oxaliplatin
  Other Names: OXA
Drug: Capecitabine
  Other Names: CAPE
Radiation: intensity modulated radiotherapy
  Other Names: IMRT
Procedure: DRE-Endoscopy-MRI-CEA
Procedure: Nonoperative Management
  Other Names: NOM
  Groups: Group A:Clinical complete response (cCR); Group B:Near-cCR
Procedure: Local Excision
  Other Names: LE
  Groups: Group B:Near-cCR
Procedure: Total Mesorectal Excision
  Other Names: TME
  Groups: Group C:Residual tumor
Behavioral: Quality of Life Questionnaires

SUMMARY:
This study is designed to test the efficacy of tailored operative or non-operative management (NOM) for MRI defined low-risk rectal cancer following neoadjuvant intensity modulated radiotherapy with concurrent capecitabine plus consolidation CapeOX. The main purpose of this study is to increase organ-preservation rate for low-risk rectal cancer patients.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiotherapy (nCRT), total mesorectal excision and adjuvant chemotherapy comprise the standard treatment for locally advanced rectal cancer, following which 15-30% patients achieved pathological complete response need to receive the removal of rectum without residual tumor and suffer significant functional impairment even after sphincter preservation. Adjuvant chemotherapy is also questioned for its benefit for prolonged survival through the data from various studies. More evidence demonstrated that organ-preservation (e.g. non-operative management or local excision) for patients with clinical complete response (cCR) or near-cCR following nCRT had similar survival when compared with those received standard care.

This study is designed to investigate the efficacy of neoadjuvant intensity modulated nCRT with concurrent capecitabine plus consolidation CapeOX for T2/DWI/Enhanced MRI defined cT2-T3b mid-low rectal cancer without threatening mesorectal fascia or extramural vascular invasion (EMVI) or mrN2 disease.

According to the response to treatment evaluated by multi-modal assessment including digital exam, T2/DWI/Enhanced MRI, endoscopy and serum CEA test, patients will receive tailored operative management like local excision or total mesorectal excision, or non-operative management. Intention to treatment was also allowed in this study.

Firstly, the investigators will observe the organ preservation rate at 2 years. Endpoints for organ-preservation like non-regrowth DFS, stoma-free survival and other conventional survival outcomes (DFS, OS) would be further collected. The short-term and long-term QoL will be measured in all patients.

. Our baseline data showed the 48% of locally advanced rectal cancers could be downstaged to stage ypT0-2N0 following IMRT with concurrent capecitabine. We hypothesize that at least 24% of rectal cancers could be candidates for LE or NOM after IMRT and the rectum preservation rate will increase to 40% in low-risk rectal cancers by LE or NOM following IMRT plus consolidation CapeOX at 2 years. As a superiority design, this study need to recruit 64 patients to test this hypothesis, with 85% power (exact binomial test for proportions, alpha = 5 %, one-sided), If the number of responses is 22 or more, the hypothesis that P <= 0.240 is rejected. We anticipate about 10 % loss to follow-up, so we will recruit an additional 8 patients and the study will recruit 72 patients in all.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤85 years
* ECOG Performance status 0-1
* Histologically confirmed diagnosis of adenocarcinoma of the rectum, with tumor differentiation Grade 1-3
* The distance from down verge of tumor to anal-rectal junction (ARJ) ≤8cm based on MRI, or ≤12cm based on sigmoidoscopy;
* Clinical Stage T2 or T3a or T3b and EMVI (-) and MRF (-) and extra-mesorectal metastatic lymph node (-) based on MRI
* No evidence of distant metastases
* No prior pelvic radiation therapy
* No prior chemotherapy or surgery for rectal cancer
* No active infections requiring systemic antibiotic treatment
* ANC > 1.5 cells/mm3, HGB > 10.0 g/dL, PLT > 100,000/mm3, total bilirubin ≤ 1.5 x ULN, AST≤ 3 x ULN, ALT ≤ 3 x ULN.
* Patients must read, agree to, and sign a statement of Informed Consent prior to participation in this study.

Exclusion Criteria:

* Recurrent rectal cancer
* Primary unresectable rectal cancer. A tumor is considered unresectable when invading adjacent organs and an en-bloc resection will not achieve negative margins.
* Creatinine level greater than 1.5 times the upper limit of normal.
* Patients who have received prior pelvic radiotherapy.
* Patients who are unable to undergo an MRI.
* Patients with a history of a prior malignancy within the past 5 years, except for well treated basal cell cancer, squamous cell skin cancer, breast cancer, thyroid cancer or small renal cancer, and with DFS >5 years.
* Patients with a history of any arterial thrombotic event within the past 6 months. This includes angina (stable or unstable), MI, TIA, or CVA.
* Other Anticancer or Experimental Therapy.
* Women who are pregnant or breast-feeding.
* Patients with any other concurrent medical or psychiatric condition or disease which would make them inappropriate candidates for entry into this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patient who receives primary care in Beijing Cancer Hospital will be selected as the candidate for this study.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2016-08; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Organ preservation rate | 3 years
  The rate of organ preservation will be defined as the percentage of patients who achieve cCR or near-cCR after neoadjuvant treatment followed by local excision or non-operative management (NOM). The time of organ preservation will be measured from the initiation of treatment.

SECONDARY OUTCOMES:
Rate of non-regrowth disease-free survival (NR-DFS) | 3 years
  NR-DFS will be defined as the length of time after treatment until death (any cause), tumor relapse including local pelvic recurrence following TME or local resection and any distant metastasis during or after treatment. Surgical salvageable local regrowth occurs in non-operative management will not be defined as tumor relapse.
Stoma-free survival | 3 years
  Stoma-free survival will be defined as the length of time in which patients live with a temporary or permanent stoma and be measured from the initiation of treatment. Events for stoma-free survival are temporary or permanent stoma or death (any cause). Temporary ileostomy-free survival or colostomy-free survival will also be calculated.
Major adverse events | 3 years
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) | Time0: before neoadjuvant treatment; Time1: at 4 months after the completion of neoadjuvant radiation; Time2: 12 months after Time1; Time3: 24 months after Time1; Time4: 36 months after Time1
  EORTC QLQ-C30 (Aaronson et al., 1993). The questionnaire assesses health status and quality of life of cancer patients using 30 items grouped in one global scale, five multi-item functioning scales, three symptom scales and six single symptom items.
  The items are scored on a four-point Likert scale with higher scores indicating a better level of functioning or a higher level of symptoms. The validity and reliability of the Mandarin versions of the questionnaire have been established.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Colorectal Cancer Module 29 (EORTC QLQ-CR29) | Time0: before neoadjuvant treatment; Time1: at 4 months after the completion of neoadjuvant radiation; Time2: 12 months after Time1; Time3: 24 months after Time1; Time4: 36 months after Time1
  EORTC QLQ-CR29 (Whistance et al., 2009). The questionnaire measures health-related quality of life in patients with colorectal cancer, using 29 items grouped in four functional scale and 18 symptom scale The items are scored on a four-point Likert scale with higher scores indicating a better level of functioning or a higher level of symptoms. The validity and reliability of the Mandarin versions of the questionnaire have been established.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang L, Zhang XY, Zhao YM, Li SJ, Li ZW, Sun YS, Wang WH, Wu AW; Rectal Cancer Cooperative Group of Peking University Cancer Hospital. Intentional Watch and Wait or Organ Preservation Surgery Following Neoadjuvant Chemoradiotherapy Plus Consolidation CAPEOX for MRI-defined Low-risk Rectal Cancer: Findings From a Prospective Phase 2 Trial (PKUCH-R01 Trial, NCT02860234). Ann Surg. 2023 Apr 1;277(4):647-654. doi: 10.1097/SLA.0000000000005507. Epub 2022 Jun 29. PMID 35766394